CLINICAL TRIAL: NCT03890718
Title: Topography Versus Non-Topography-Guided Photorefractive Keratectomy With Corneal Cross-Linking Variations in Keratoconus
Brief Title: Topography Versus Non-Topography-Guided PRK With CXL in Keratoconus
Acronym: keratoconus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Principal Investigator, farinaz doroodgar, Ophthalmologist, Shahid Beheshti University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ShaheidBU
Record Dates: First submitted 2019-03-25; First posted 2019-03-26 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-01

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus | interventions — Photorefractive Keratectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Photorefractive keratectomy in mile keratoconus (Experimental): Photorefractive keratectomy in mile keratoconus type of corneal surface ablation in for correct refractive error
  Interventions: Procedure: Photorefractive keratectomy in mile keratoconus

INTERVENTIONS:
Procedure: Photorefractive keratectomy in mile keratoconus — Topo-guided photorefractive keratectomy will be performed using an excimer laser (Allegretto Wave Topolyzer, Alcon, Inc.) with a 6 mm optical area and a transition area of 2 mm in all eyes. At that point, the partial topography-guided photorefractive keratectomy laser treatment will be finished. The arrangement will be to treat 70% of the cylindrical and spherical part to not surpass 50μm of stromal expulsion. The estimation of 50μm as the most extreme removal depth recommended by Kanellopoulos in Athens protocol will be chosen
  Other Names: Advance surface abelation in mild keratoconus

SUMMARY:
To our knowledge, this study is one of the first to compare the visual results of non-topography-guided and topography-guided photorefractive keratectomy (PRK) applying sequential and simultaneous corneal cross-linking (CXL) treatment for keratoconus. Considering recent advances in cross-linking and imaging in keratoconus, the outcomes of this study can lead us to several non-invasive algorithm management options.

DETAILED DESCRIPTION:
Interventional and comparative prospective study: Sixty-nine eyes (38 patients) suffering from keratoconus (stages 1-2 Amsler-Krumeich classification) were divided into four groups. The four groups underwent topography- and non-topography-guided PRK with sequential and simultaneous CXL. The main outcome measures were pre- and postoperative uncorrected distance visual acuity (UDVA), best corrected distance visual acuity (CDVA), manifest refraction, contrast sensitivity, and keratometry.

ELIGIBILITY:
Inclusion criteria

* age 34 (range from 34 to 41)
* stable corneal topography and refraction for at least six months
* estimated residual bed thickness of >410 µm

Exclusion

* presence of macular or retinal disease,
* dry eye
* history of recurrent corneal erosions
* anterior segment abnormalities
* unstable refractive error
* post-surgically residual stromal bed thickness of under 350 mm
* autoimmune disease
* collagen vascular disease
* immunosuppressive therapy or current use of systemic corticosteroids
* diabetes mellitus
* pregnancy
* lactation

Ages: 34 Years to 41 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2017-03-30 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
visual acuity | 3 months
  Visual acuity (VA) commonly refers to the clarity of vision

OTHER OUTCOMES:
Aberrometry properties by iTrace Ray-tracing aberrometry | 3 year
  Optical aberrations are a major cause for poor quality of vision. It occurs when light from one point, after transmission through an optical system, does not converge to or diverge from a single point. Any deviation of the optical system from paraxial optics results in aberrations. In the eye, the various refracting surfaces like tear film, cornea and lens are primarily responsible for inducing ocular aberrations. The difference in shape of the wave-front entering the eye and that exiting the eye defines the type of aberration. The ocular aberrations are classified into lower order aberration (LOA) (zero order- piston; first order- horizontal and vertical tilt; second order- spherical defocus and astigmatism) and higher order aberrations (HOA) (third order - coma and trefoil; fourth order - quatrefoil, secondary astigmatism and spherical aberrations; fifth order - pentafoil; sixth order - hexafoil).

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Alio, MD,PhD, Study Chair — Division of Ophthalmology, Universidad Miguel Hernández, Alicante, Spain
Locations (1):
- Farideh Doroodgar, Tehran, Iran